CLINICAL TRIAL: NCT01387750
Title: Evaluating the Efficacy, Tolerance and Acceptability of a Mentholated Cream Containing Oxygenated Glycerol Triesters (OGT) on Acute Pain in Subjects Suffering From a Recent Inflammation of the Muscles and/or Joints
Brief Title: Mentholated Cream Containing Oxygenated Glycerol Triesters on Acute Pain of the Muscles and Joints
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Collaborators: Laboratories Carilene (Unknown)
Responsible Party: Barry T. Reece, MS, MBA, Reliance Clinical Trial Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCTS2223
Record Dates: First submitted 2011-06-30; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Pain; Analgesics
Keywords: Acute Pain; Musculoskeletal Pain; Topical Analgesic
MeSH Terms: conditions — Pain; Acute Pain; Musculoskeletal Pain | interventions — UDP-N-acetylglucosamine-peptide beta-N-acetylglucosaminyltransferase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mentholated Cream (Placebo Comparator)
  Interventions: Other: Mentholated Cream
- Mentholated Cream with OGT (Active Comparator)
  Interventions: Other: Mentholated Cream with OGT

INTERVENTIONS:
Other: Mentholated Cream — A topical cream containing menthol without the addition of the oxygenated glycerol triesters.
  Arms: Mentholated Cream
Other: Mentholated Cream with OGT — A Topical Cream that contained both menthol and oxygenated glycerol triesters.
  Arms: Mentholated Cream with OGT

SUMMARY:
A single center trial to evaluate the efficacy, tolerance, and acceptability of Oxygenated Glycerol Triesters (OGT) mentholated cream on acute musculoskeletal pain in normal healthy adult volunteers suffering from a recent inflammation of muscles and joints. Patient who met eligibility requirements were instructed to identify one area on their body where they were experiencing the most acute musculoskeletal pain/discomfort. Patients were provided with visual analog scales in order to quantify their pain. Patients either received mentholated cream with or without OGT and instructed to rub on the identified site 3 times a day for 7 days. Pain and other observations were written in a diary for each day.

ELIGIBILITY:
Inclusion Criteria:

1. Were males and females between the ages of 18 and 75, in good general health (no physical required but subjects did fill out a medical history questionnaire)
2. Were individuals free of any systemic or dermatological disorder including a known history of allergies or other medical conditions which, in the opinion of the investigator, might have interfered with the conduct of the study, interpretation of results or increased the risk of adverse reactions;
3. Were individuals that had recently (< three months) started to suffer from acute musculoskeletal pain (i.e. arthritis, simple back pain, muscle strains);
4. Agreed to stop any anti-inflammatory or analgesic medications two days prior to starting the study;
5. Had the ability to complete the course of the study and to comply with instructions;
6. Agreed not to use or introduce any new personal care products (including cosmetics, skin care, hand care, body care, hair care, personal hygiene, etc.) into their normal regimen during the course of the study;
7. Agreed to avoid sun exposure during the course of the study;
8. Were females that were surgically sterile, post-menopausal or using an acceptable method of birth control; and
9. Were able to read, understand and provide written informed consent.

Exclusion Criteria:

1. Were individuals with any visible skin disease or skin condition (e.g., eczema), which might have interfered with the evaluations;
2. Were individuals with excessive dryness or redness at the sites of application;
3. Were individuals who suffered from chronic and/or severe musculoskeletal pain;
4. Were individuals with a known hypersensitivity to topical analgesics or other pain relieving products;
5. Were females who were pregnant, planning a pregnancy or nursing a child;
6. Were individuals who were participating, or had participated, on a clinical study involving the body (exclusive of the face) within 28 days prior to study initiation;
7. Were individuals who had psoriasis;
8. Were individuals currently under treatment for asthma or diabetes (insulin-dependent only);
9. Were individuals with active atopic dermatitis/eczema at the test sites;
10. Were individuals taking prescription or over-the-counter anti-inflammatory medications, non- steroidal anti-inflammatory drugs and topical, oral and systemic steroids; and
11. Were individuals with known allergies to any of the components of the test articles.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Severity of Pain
  Patients were instructed to identify one area on their body where they were experiencing the most acute musculoskeletal pain/discomfort.

SECONDARY OUTCOMES:
Limitation of Activity
  How limited patient activities were due to the pain associated with the area of interest.
Evaluation of the mobility of the painful joint/muscle
  Patient assessed how mobile their joints/muscles were within the area of interest.
Skin Toxicity
  Tolerability was assessed from Redness and Dryness VAS recorded by the clinical evaluator. No formal safety testing was performed in this study; however anecdotal information (stinging, burning, itching, etc.) was captured on the subjects' diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Barry T Reece, MS, MBA, Principal Investigator — RCTS, Inc.; Jessica Williams, BS, Study Director — RCTS, Inc.